CLINICAL TRIAL: NCT03691896
Title: The Impact of the Dose of Vitamin D (vitD) on the Metabolism of ca, p and Concentrations of 25OHD, Bone Status and Development of Premature Infants up to 2 Years of Age. Prospective, Randomized, Clinical Study
Brief Title: Calcium (ca),Phosphorus( P) and 25-hydroxyvitamin D(25OHD)] in Infants Born ≤ 32 PMA Gestational Weeks (GA)
Acronym: Ca-P
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Maria Wilinska, Head Of Neonatology, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 501-1-13-15-16
Record Dates: First submitted 2016-06-18; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Infant, Premature, Diseases
Keywords: premature; osteopenia; Vit. D; LBW (low birth weight); 25OHD
MeSH Terms: conditions — Infant, Premature, Diseases; Premature Birth; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lower dose (Experimental): cholecalciferol 400UNT, oral solution
  Interventions: Dietary Supplement: Cholecalciferol 400
- Middle dose (Active Comparator): cholecalciferol 800UNT, oral solution
  Interventions: Dietary Supplement: Cholecalciferol 800
- Higher dose (Experimental): cholecalciferol 1200UNT, oral solution,
  Interventions: Drug: Cholecalciferol 1200

INTERVENTIONS:
Dietary Supplement: Cholecalciferol 400 — dose 400 UNT/day for 12 months
  Other Names: vit D
  Arms: Lower dose
Dietary Supplement: Cholecalciferol 800 — dose 800 UNT/day for 12 months
  Other Names: vit D
  Arms: Middle dose
Drug: Cholecalciferol 1200 — dose 1200 UNT/day for 12 months
  Other Names: vit D
  Arms: Higher dose

SUMMARY:
It has not yet been established the optimal dose of vit. D for preterm infants in Poland. It is not known what dose of vit. D will provide the correct concentration of vit. D and the optimal development of the skeleton of the premature.

The study will try to determine the optimal supplementation of vitamin D and the supply of Ca and P for normal growth and development of a child born prematurely.

In addition, the investigators will evaluate any risk factors for deficiency and excess of vitamin D and the consequences of its deficiency and overdose. Simultaneously the study would make possible the determination of an optimal schedule for controlling the Ca-P levels in the group of the youngest infants born prematurely. In addition, the study will assess the relationship between maternal and newborn vitamin D resources right after birth, and the incidence of vitamin D deficiency in infants born prematurely. Preterm infants will be randomized in 3 groups assigned to different doses of vit. D. The study will investigate the metabolism of calcium, phosphorus, the health of bones and development of the premature babies till the age of 2.

DETAILED DESCRIPTION:
The participants of the study will be prematures, born ≤32 GA, hospitalized in the Department of Neonatology, in the neonatal intensive care unit. Hospitalized patients who meet the inclusion criteria will be randomized in 3 groups assigned to different doses of vit. D (400, 800 or 1200 units(UNT) of vitamin D).

At defined age points of postnatal life, parameters of calcium and phosphorus metabolism and vitamin D level will be tested, along with the health of bones, health status and development.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≤32 weeks at birth
* hospitalization in the department no later than at the age of 7 days (for infants born outside the center)
* No birth defects or diseases permanently affecting the ability to accept enteral feeding
* Anticipated possibility of continuous monitoring of the course of treatment in hospital until discharge
* Consent of Parents / legal guardians for the participation in the study.

Exclusion criteria

* gestational age> 32 weeks at birth
* the beginning of hospitalization in the department later than the age of 7 days (for infants born outside the center)
* presence of congenital defects or diseases permanently affecting the ability to accept enteral feeding (e.g.oesophageal atresia, anal atresia, congenital umbilical hernia, gastroschisis, syndromes genetically determined)
* significant interruption (> 1 week) of the hospitalization in the center
* lack of consent of the Parents / legal guardians to participation in the study

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Serum 25OHD levels in cord blood in Polish preterm infants | day of labour
  assessment of 25OH D levels in children deficiency: <10ng/ml, insufficient level: 10-30ng/ml, sufficient level: 30-50ng/ml

SECONDARY OUTCOMES:
Impact of supplementation of Vit. D during pregnancy on 25OHD serum level in Polish mothers | day of labour
  assessment of 25OH D levels in mothers deficiency: <10ng/ml, insufficient level: 10-30ng/ml, sufficient level: 30-50ng/ml
Impact of dosage of Vit D3 (400/800/1200 UNT per day) on serum 25OH D levels in preterm children | 4,8,12 weeks of life,1 and 2 years of age
  assessment of serum 25OH D levels in children deficiency: <10ng/ml, insufficient level: 10-30ng/ml, sufficient level: 30-50ng/ml; high level > 60ng/ml, toxic level > 100ng/ml
Impact of dosage of Vit D3 (400/800/1200 UNT /per day) on Ca serum levels | 4,8,12 weeks of life,1 and 2 years of age
  assessment of Ca serum levels in children
Impact of dosage of Vit D3 (400/800/1200 UNT /per day) on P serum levels | 4,8,12 weeks of life,1 and 2 years of age
  assessment of P serum levels in children
Impact of dosage of Vit D3 (400/800/1200 UNT /per day) on urinary Ca excretion | 4,8,12 weeks of life,1 and 2 years of age
  assessment of urinary calcium/creatinine index
Impact of dosage of Vit D3 (400/800/1200 UNT /per day) on urinary P excretion | 4,8,12 weeks of life,1 and 2 years of age
  assessment of urinary P/creatinine index (mg/mg)
impact of total annual Vit D3 dose and bone calcification in children | average of 1 and 2 years of age
  assessment of bone status :Densitometry (DEXA)
correlation of cord blood 25OHD level and GA | 1st day of life
  birth <24 GA, 24-28GA, 28-32GA
impact of cord blood 25OHD level on birth weight | 1st day of life of age
  assessment of percentile of birth weight (Fenton 2013) hypotrophy <3p, eutrophy 3-97p, hypertrophy >97p

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Zarlenga, MD, Principal Investigator — Mc postgraduate SPSK im prof.W.Orłowskiego Warszawa; Maria Wilińska, DSc, Study Chair — Mc postgraduate SPSK im prof.W.Orłowskiego Warszawa; Ewa Głuszczak-Idziakowska, PhD, Principal Investigator — Mc postgraduate SPSK im prof.W.Orłowskiego Warszawa
Locations (1):
- SPSK im. prof. W.Orłowskiego CMKP Neonatology Departament, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bodnar LM, Klebanoff MA, Gernand AD, Platt RW, Parks WT, Catov JM, Simhan HN. Maternal vitamin D status and spontaneous preterm birth by placental histology in the US Collaborative Perinatal Project. Am J Epidemiol. 2014 Jan 15;179(2):168-76. doi: 10.1093/aje/kwt237. Epub 2013 Oct 11. PMID 24124195
- [Background] Monangi N, Slaughter JL, Dawodu A, Smith C, Akinbi HT. Vitamin D status of early preterm infants and the effects of vitamin D intake during hospital stay. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F166-8. doi: 10.1136/archdischild-2013-303999. Epub 2013 Jul 13. PMID 23852093
- [Background] Natarajan CK, Sankar MJ, Agarwal R, Pratap OT, Jain V, Gupta N, Gupta AK, Deorari AK, Paul VK, Sreenivas V. Trial of daily vitamin D supplementation in preterm infants. Pediatrics. 2014 Mar;133(3):e628-34. doi: 10.1542/peds.2012-3395. Epub 2014 Feb 10. PMID 24515510
- [Background] van de Lagemaat M, Rotteveel J, Schaafsma A, van Weissenbruch MM, Lafeber HN. Higher vitamin D intake in preterm infants fed an isocaloric, protein- and mineral-enriched postdischarge formula is associated with increased bone accretion. J Nutr. 2013 Sep;143(9):1439-44. doi: 10.3945/jn.113.178111. Epub 2013 Jul 31. PMID 23902955
- [Background] Schanler RJ, Burns PA, Abrams SA, Garza C. Bone mineralization outcomes in human milk-fed preterm infants. Pediatr Res. 1992 Jun;31(6):583-6. doi: 10.1203/00006450-199206000-00009. PMID 1635820
- [Background] Kislal FM, Dilmen U. Effect of different doses of vitamin D on osteocalcin and deoxypyridinoline in preterm infants. Pediatr Int. 2008 Apr;50(2):204-7. doi: 10.1111/j.1442-200X.2008.02553.x. PMID 18353060
- [Background] Christmann V, de Grauw AM, Visser R, Matthijsse RP, van Goudoever JB, van Heijst AF. Early postnatal calcium and phosphorus metabolism in preterm infants. J Pediatr Gastroenterol Nutr. 2014 Apr;58(4):398-403. doi: 10.1097/MPG.0000000000000251. PMID 24253367
- [Background] Backstrom MC, Maki R, Kuusela AL, Sievanen H, Koivisto AM, Koskinen M, Ikonen RS, Maki M. The long-term effect of early mineral, vitamin D, and breast milk intake on bone mineral status in 9- to 11-year-old children born prematurely. J Pediatr Gastroenterol Nutr. 1999 Nov;29(5):575-82. doi: 10.1097/00005176-199911000-00019. PMID 10554126
- [Background] Fewtrell MS, Prentice A, Jones SC, Bishop NJ, Stirling D, Buffenstein R, Lunt M, Cole TJ, Lucas A. Bone mineralization and turnover in preterm infants at 8-12 years of age: the effect of early diet. J Bone Miner Res. 1999 May;14(5):810-20. doi: 10.1359/jbmr.1999.14.5.810. PMID 10320530
- [Background] McCarthy RA, McKenna MJ, Oyefeso O, Uduma O, Murray BF, Brady JJ, Kilbane MT, Murphy JF, Twomey A, O' Donnell CP, Murphy NP, Molloy EJ. Vitamin D nutritional status in preterm infants and response to supplementation. Br J Nutr. 2013 Jul 14;110(1):156-63. doi: 10.1017/S0007114512004722. Epub 2012 Nov 27. PMID 23182428